CLINICAL TRIAL: NCT03456934
Title: Lower Protein Intake and Long-term Risk of Obesity and Cardiovascular Disease: A Multi-centred, Randomised, Controlled Trial
Brief Title: Lower Protein Intake and Long-term Risk of Obesity and Cardiovascular Disease
Acronym: BabyGrowth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15.09.INF
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Infant Formula; Growth
Keywords: Protein requirements; Adiposity; Body composition; Cardiovascular health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind with nonrandomized breast-fed reference group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Modified infant formula given from 3 to 12 months of age, as per standard requirement.
  Interventions: Other: Modified infant formula
- Control Group (Active Comparator): Standard infant formula given from 3 to 12 months of age, as per standard requirement.
  Interventions: Other: Standard infant formula
- Breast-fed Reference Group (No Intervention): Non-randomized infants who are predominantly breast-fed at time of enrollment.

INTERVENTIONS:
Other: Modified infant formula — Test formula with lower protein content than standard formula
  Arms: Experimental Group
Other: Standard infant formula — Standard infant formula
  Arms: Control Group

SUMMARY:
The primary objective of this study is to investigate if consumption of lower protein formula can slow the rate of weight gain of formula-fed infants between 3 and 12 months of age. Secondary objectives include investigation into whether infant nutrition and growth have an impact on later risk of obesity and cardiovascular disease.

DETAILED DESCRIPTION:
Obesity and its cardiovascular consequences are the most important causes of morbidity and mortality worldwide. Breastfed infants have been shown to have less cardiovascular risk factors in adulthood, which can be partially explained by their slower growth compared to formula fed infants. The primary objective of this study is to investigate if consumption of lower protein formula can slow the rate of weight gain of formula-fed infants between 3 and 12 months of age. Secondary objectives include investigation into whether infant nutrition and growth have an impact on later risk of obesity and atherosclerotic cardiovascular disease (CVD), the critical windows for these programming effects, and the mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infant
* Infant is aged 14 weeks (+/- 1 week)
* Infant is exclusively formula feeding or predominantly breast-feeding at age 14 weeks

Exclusion Criteria:

* Any adverse maternal, fetal or infant medical history that may have effects on growth and/or development
* Infant born with congenital disease or malformation affecting growth and/or development
* Food allergy to any trial products (e.g. milk, soy)

Ages: 13 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Infant weight gain | Between ages 14 weeks (+/- 1 week) and 12 months (+/- 2 weeks)
  Rate of weight gain (g/d)

SECONDARY OUTCOMES:
Body mass index (BMI)-for-age Z-score | Age 2 years (+/- 1 month)
  Based on World Health Organization (WHO) growth standards
Height-for-age Z-score | Age 2 years (+/- 1 month)
  Based on WHO growth standards
Adiposity | Age 2 years (+/- 1 month)
  Sum of 4 skinfolds (triceps, biceps, sub-scapular, supra-iliac)
Fat mass | Age 2 years (+/- 1 month)
  Deuterium dilution (assessed in subset)

OTHER OUTCOMES:
Infant weight gain | Between 6 and 12 months
  Rate of weight gain (g/d)
Weight | Ages 4, 5, 6, 12 and 24 months
  Body weight (kg)
Length or height | Ages 4, 5, 6, 12 and 24 months
  Length or height (cm)
Head circumference | Ages 4, 5, 6, 12 and 24 months
  Head circumference (cm)
Body mass index | Ages 6, 12 and 24 months
  Weight and length or height will be combined to report BMI in kg/m^2
Weight-for-age Z-score | Ages 14 weeks and 4, 5, 6, 12 and 24 months
  Based on WHO growth standards
Weight-for-length Z-score | Ages 14 weeks and 4, 5, 6, 12 and 24 months
  Based on WHO growth standards
Height-for-age Z-score | Ages 14 weeks and 4, 5, 6, and 12 months
  Based on WHO growth standards
BMI-for-age Z-score | Ages 14 weeks and 4, 5, 6, and 12 months
  Based on WHO growth standards
Adverse events | Ages 14 weeks and 4, 5, 6, 9, 12 and 24 months
  Safety
Feeding intake | Ages 14 weeks and 4, 5, 6, and 12 months
  Infant feeding questionnaire
Feeding tolerance | Ages 14 weeks and 4, 5, 6, and 12 months
  GI symptom and stool pattern questionnaire
Metabolic markers of cardiovascular health | Ages 6 and 12 months
  Blood sample (in a subset)
Blood pressure | At age 12 and 24 months
  Systolic and diastolic blood pressure (in a subset)
Appetite and feeding / eating behavior | Ages 14 weeks and 4, 5, 6, and 24 months
  Baby and Children's Eating Behavior Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Atul Singhal, MD, Principal Investigator — Childhood Nutrition Research Centre, University College London, Institute of Child Health
Locations (1):
- UCL Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831